CLINICAL TRIAL: NCT05019118
Title: Dietary Intervention With Únicla Dairy Products, Naturally Enriched With Selenium and Omega-3 Fatty Acids, May Improve Thyroid-stimulating Hormone (TSH) Levels in Women With Subclinical Hypothyroidism
Brief Title: Dietary Intervention With Únicla Dairy Products (DANTIAN)
Acronym: DANTIAN
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cooperativas Lacteas Unidas (Industry)
Collaborators: Galician South Health Research Institute (Network)
Responsible Party: Principal Investigator, María Reyes Pérez Fernández, PhD Clinical Professor, Galician South Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CLUN-20191005
Record Dates: First submitted 2021-08-13; First posted 2021-08-24 (Actual); Last update posted 2021-08-24 (Actual); Status verified 2021-08

CONDITIONS: Subclinical Hypothyroidism
Keywords: Hypothyroidism; selenium; women
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Intervention Model Description: Randomized, masked and controlled nutritional intervention study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The masking process will be triple blind, that is, both the participating women, the research staff (including those in charge of delivering the products and the one who performs and interprets the measurements), as well as the analyst, won't know at any time what group belong to patients. All the products in the study (Únicla dairy) as well as their respective placebos (conventional FEIRACO equivalent products) will maintain a similar format and labeling, with the organoleptic characteristics of dairy products being very similar. Masking will be opened at the time that the last data interpretation of the last subject included was made and before starting the statistical analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention/treatment (Experimental): Dairy foods made with UNICLA milk Participants (n = 45) ingested UNICLA milk and dairy products (yogurt and cheese) for three months.
  UNICLA milk is characterised by an improved nutritional composition, obtained by modifying cow's diet, feeeding the dairy cows with a sufficient and balanced ration, which recreates the fatty acid profile of the spring.
  This ration includes pastures, high-quality forages and, among other components, a significant amount of flax seeds, which constitute a source of unsaturated fatty acids such as omega-3 and selenised yeast, as a source of organic selenium.
  Consequently, UNICLA milk and dairy products are naturally enriched in selenium and ω-3 PUFA.
  The daily intake reflects the usual consumption habits, being the recommended amounts of 200 ml of milk and 125 g of yogurt per day and 400g of fresh cheese per week
  Interventions: Other: Experimental milk; Other: Experimental yogur; Other: Experimental fresh cheese
- Conventional milk (Placebo Comparator): Participants (n = 45) ingest milk and conventional dairy products daily for 3 months.
  Daily intake reflects usual dairy consumption habits in "real life" conditions, without forcing or inducing increased consumption. Therefore, the recommended amounts are 200 ml of milk and 125 g of yogurt per day and 400 g of fresh cheese per week
  Interventions: Other: Placebo milk; Other: Placebo yogur; Other: Placebo fresh cheese

INTERVENTIONS:
Other: Experimental milk — UNICLA milk naturally enriched in selenium and omega-3.
  Other Names: ÚNICLA milk
  Arms: Intervention/treatment
Other: Experimental yogur — UNICLA yogur naturally enriched in selenium and omega-3.
  Other Names: ÚNICLA yogur
  Arms: Intervention/treatment
Other: Experimental fresh cheese — UNICLA fresh cheese naturally enriched in selenium and omega-3.
  Other Names: ÚNICLA fresh cheese
  Arms: Intervention/treatment
Other: Placebo milk — Conventional milk
  Other Names: Conventional milk
  Arms: Conventional milk
Other: Placebo yogur — Conventional yogur
  Other Names: Conventional yogur
  Arms: Conventional milk
Other: Placebo fresh cheese — Conventional fresh cheese
  Other Names: Conventional fresh cheese
  Arms: Conventional milk

SUMMARY:
Dietary intervention with Únicla dairy products, naturally enriched with selenium and omega-3 fatty acids, may improve thyroid-stimulating hormone (TSH) levels in women with subclinical hypothyroidism

DETAILED DESCRIPTION:
To analyze in women diagnosed with subclinical hypothyroidism, the effects of consumption of dairy products rich in selenium and omega-3 on symptoms related to thyroid disease and blood lipid profile, inflammatory response, and fatty acid levels in the red blood cell membrane among others.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of subclinical hypothyroidism
* TSH levels between 3 and 10 mIU / L
* Normal levels of free triiodothyronine ( T3) and free thyroxine (T4)
* Without previous or current treatment with levothyroxine

Exclusion Criteria:

* Thyroid surgery or reception of radioactive iodine in a previous period of 12 months
* History of cardiovascular disease and / or thrombosis
* Established diagnosis or clinical suspicion of kidney or liver failure, chronic infections, blood diseases, type I diabetes and type II diabetes
* Drug treatments that affect thyroid function (corticosteroids, amiodarone, propranolol, lithium)
* Statin treatment and / or hormone replacement therapy
* Adjuvant treatment with trace elements, vitamins or antidepressant and antipsychotic drugs
* Hospitalization for serious illness or elective surgery in the past 4 weeks
* Diseases and / or treatments that affect intestinal absorption (proton pump inhibitors)
* Pregnant, planning to become pregnant or breastfeeding women
* Consumption of ω-3 PUFA type food supplements
* Intolerance and / or allergy to lactose and / or cow's milk proteins
* Any pathology that requires close control, advises against their participation or there is an inability to move independently
* Habitual residence outside the study's influence area
* Participation in another clinical trial with drugs, or in other experimental studies
* Refuse to sign the informed consent

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2021-09-06 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with changes in thyroid function | 3 months
  thyroid stimulating hormone blood level

SECONDARY OUTCOMES:
HDL level | 3 months
  high density lipoproteins blood level
selenium | 3 months
  selenium blood level
IL-6 | 3 months
  Interleukina-6 blood level
Fecal calprotectin | 3 months
  Fecal calprotectin feces level

CONTACTS AND LOCATIONS:
Overall Officials: Maria Reyes Pérez- Fernández, PhD, Principal Investigator — Galicia sur sanitary research institute
Locations (1):
- Nursing University School of Ourense, Ourense, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Roibas L, Martinez I, Goris A, Barreiro R, Hospido A. An analysis on how switching to a more balanced and naturally improved milk would affect consumer health and the environment. Sci Total Environ. 2016 Oct 1;566-567:685-697. doi: 10.1016/j.scitotenv.2016.05.141. Epub 2016 May 27. PMID 27239712
- [Background] Muniz-Naveiro O, Dominguez-Gonzalez R, Bermejo-Barrera A, Cocho de Juan JA, Fraga Bermudez JM, Goris Pereiras A, Lopez Santamarina A, Martinez Lede I, Valledor Puente J, Fernandez-Couto Gomez L, Bermejo-Barrera P. Selenium content and distribution in cow's milk supplemented with two dietary selenium sources. J Agric Food Chem. 2005 Dec 14;53(25):9817-22. doi: 10.1021/jf050155w. PMID 16332137
- See also: Article preprint magazine Nutrition Hospitalaria — https://www.google.com/search?q=Efectos+de+la+ingesta+de+l%C3%A1cteos+enriquecidos+de+forma+natural+con+selenio+y+omega-3+en+una+muestra+de+mujeres+postmenop%C3%A1usicas+con+s%C3%ADndrome+metab%C3%B3lico%3A+un+ensayo+cl%C3%ADnico+aleatorizado+triple+ciego+y+controlado+con+placebo&oq=Efectos+de+la+ingesta+de+l%C3%A1cteos+enriquecidos+de+forma+natural+con+selenio+y+omega-3+en+una+muestra+de+mujeres+postmenop%C3%A1usicas+con+s%C3%ADndrome+metab%C3%B3lico%3A+un+ensayo+cl%C3%ADnico+aleatorizado+triple+ciego+y+controlado+con+placebo&aqs=chrome..69i57.5124j0j4&sourceid=chrome&ie=UTF-8